CLINICAL TRIAL: NCT03749070
Title: Efficacy of Silymarin in Patients With Non-alcoholic Fatty Liver Disease - The SILIVER Trial: Randomized Clinical Trial
Brief Title: Efficacy of Silymarin in Patients With Non-alcoholic Fatty Liver Disease - The SILIVER Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Camila Ribeiro de Avelar (Other)
Responsible Party: Sponsor-Investigator, Camila Ribeiro de Avelar, Doctor student, Hospital Universitário Professor Edgard Santos
Organization: Hospital Universitário Professor Edgard Santos (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2.635.954
Record Dates: First submitted 2018-10-28; First posted 2018-11-21 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Non-Alcoholic Fatty Liver Disease; sylimarin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Silymarin

STUDY DESIGN:
Intervention Model Description: Clinical trial, randomized, double-blind and controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silymarin (Active Comparator): Patients will receive 2 capsules containing a total of 700mg of silymarin, 8mg of vitamin E and 50mg of phosphatidylcholine, in addition to the excipient, which should be ingested daily for 12 weeks.
  Interventions: Dietary Supplement: Silymarin
- Placebo (Placebo Comparator): Patients will also receive similarly 2 capsules per day, but without the bioactive principle tested (silymarin). Therefore, the capsules in the control group will contain only 700 mg of maltodextrin, a neutral food component derived from starch, in addition to the excipient and the same amount of vitamin E and phosphatidylcholine to balance the two groups.
  Interventions: Dietary Supplement: Silymarin

INTERVENTIONS:
Dietary Supplement: Silymarin — It is a randomized, double-blind, controlled clinical trial to be performed at outpatient level. The intervention will last 12 weeks and the invited participants will be patients attended at the outpatient clinic of the Edgard Santos Hospital, which will be randomized into two groups: control and intervention. Data on laboratory and clinical markers, imaging, nutritional and dietary assessment will be collected at the beginning and end of the trial for comparison purposes.

SUMMARY:
Non-Alcoholic Fatty Liver Disease (NAFLD) is one of the most prevalent chronic liver diseases in Brazil and its treatment is still limited. Thus, this project aims to conduct a double-blind, controlled, randomized clinical trial to evaluate the effect of silymarin on laboratory markers and clinical evolution of adult patients with NAFLD treated at Edgard Santos Hospital, as well as identify the dietary pattern of these individuals.

DETAILED DESCRIPTION:
Non-Alcoholic Fatty Liver Disease (NAFLD) is one of the most prevalent chronic liver diseases in Brazil. It has a significantly increasing incidence today and is considered an important global health problem. It affects approximately 20 to 30% of the adult population and increases according to the severity of the risk factors. The diagnosis of this disease usually occurs in 10 to 20% of the non-obese individuals, 50% in the overweight and 80 to 90% in the obese, being twice as present in individuals with Metabolic Syndrome. Pharmacological treatment options for NAFLD are still limited and Silybum marianum, one of the most sought-after herbal remedies in patients with liver disease, is commonly used by patients because of the claim of the hepatoprotective effect of silymarin. Studies have demonstrated the therapeutic potential of silymarin in patients with NAFLD, but clinical trials with more judicious methodological designs is still needed to prove these effects. Thus, this project aims to evaluate the efficacy of silymarin in adult patients with NAFLD seen at the Clinic of Nutrition and Hepatology of Edgard Santos Hospital. A randomized, double-blind, controlled clinical trial lasting 12 weeks will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 20 and 60 years of age, both men and women,
* Clinical diagnosis of NAFLD, confirmed by imaging exams,

Exclusion Criteria:

* Women in the menacing period, with the exception of those who have performed definitive sterilization, such as hysterectomy or tubal ligation.
* Patients with established prior diagnosis of chronic noncommunicable disease (congestive heart failure, decompensated or severe lung disease, neoplasms, renal disease, advanced liver disease - Child Pugh C classification)
* Patients with schistosomiasis;
* Hemochromatosis
* Wilson's disease
* Viral or autoimmune hepatitis
* HIV virus carriers
* Woman who is breastfeeding
* Users of illicit drugs
* Patients with an intake of more than 20 g / day of alcohol and / or past alcoholism with abstention less than 6 months;
* Patients with ingestion of medications such as steroids, estrogens, amiodarone, warfarin, anti-convulsants, antipsychotics, tamoxifen or other chemotherapeutic agents in the last 6 months
* Patients with clinically manifest infections or inflammation, surgery, trauma or hospitalization in the last 30 days
* Chronic non-hepatic degenerative diseases (sclerosis, Parkinson's disease or Alzheimer's disease)
* Patients who do not participate in all stages of the research.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Absence or change in NAFLD degree | They will be dosed at baseline and after 12 weeks of intervention.
  Absence or change in NAFLD degree, assessed by the value of the difference in the attenuation coefficient between liver and spleen obtained by computed tomography of the upper abdomen performed at the beginning and at the end of the study.

SECONDARY OUTCOMES:
Lipid profile | They will be dosed at baseline and after 12 weeks of intervention.
  Total cholesterol (mg/dL), LDL-cholesterol (mg/dL), HDL-cholesterol (mg/dL), VLDL-cholesterol (mg/dL) and triglycerides (mg/dL) will be measured before and after the intervention.
Fasting blood glucose | They will be dosed at baseline and after 12 weeks of intervention.
  Fasting blood glucose (mg/dL) will be measured before and after the intervention.
Glycated haemoglobin | They will be dosed at baseline and after 12 weeks of intervention.
  Hb A1c (%) will be measured before and after the intervention.
Insulin | They will be dosed at baseline and after 12 weeks of intervention.
  Insulin (µU/mL) will be measured before and after the intervention.
Serum Iron | They will be dosed at baseline and after 12 weeks of intervention.
  Serum iron (mcg/dL) will be measured before and after intervention.
Transferrin saturation | They will be dosed at baseline and after 12 weeks of intervention.
  Transferrin saturation (%) will be measured before and after intervention.
Serum ferritin | They will be dosed at baseline and after 12 weeks of intervention.
  Serum ferritin will be evaluated in µg/L before and after intervention.
Hepatic transaminases | They will be dosed at baseline and after 12 weeks of intervention.
  Alanine aminotransferase (ALT) and Aspartate Aminotransferase (AST) will be evaluated in U/L before and after intervention.
gamma glutamyl transferase | They will be dosed at baseline and after 12 weeks of intervention.
  Gamma glutamyl transferase will be evaluated in U/L before and after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Camila Ribeiro de Avelar, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Avelar CR, Nunes BVC, da Silva Sassaki B, Dos Santos Vasconcelos M, de Oliveira LPM, Lyra AC, Bueno AA, de Jesus RP. Efficacy of silymarin in patients with non-alcoholic fatty liver disease - the Siliver trial: a study protocol for a randomized controlled clinical trial. Trials. 2023 Mar 10;24(1):177. doi: 10.1186/s13063-023-07210-6. PMID 36899430